CLINICAL TRIAL: NCT01232114
Title: Phase 2 Study of of a Chinese Herbal Formula Simotang Oral Liquid for the Treatment of Functional Dyspepsia
Brief Title: Safety Study of a Chinese Herbal Formula Simotang Oral Liquid for the Treatment of Functional Dyspepsia
Acronym: SMT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hunan University of Traditional Chinese Medicine (Other)
Responsible Party: Key Lab. for Chinese Internal Medicine, Hunan University of Traditional Chinese Medicine
Other Study IDs: CB523002
Record Dates: First submitted 2010-10-19; First posted 2010-11-02 (Estimated); Last update posted 2010-11-02 (Estimated); Status verified 2010-10

CONDITIONS: Functional Dyspepsia(FD) Was Studied; Effect of Simotang on FD Was Studied

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Functional dyspepsia (FD) is a common functional gastrointestinal disorder and is steadily becoming a public health problem.Simotang is a classical formula that has been used to treat gastrointestinal disorders for hundreds of years [9] and was approved as an oral liquid drug by the Chinese National Food and Drug Administration in the 1980s.In this study,patients with functional dyspepsia were divided according to the inclusive criteria into treatment group and control group randomly, who were given Simo decoction or Domperidone tablets for 14 days。And then the gastric emptying, Symptoms in plasma were observed before and after treatment in mult-center.

ELIGIBILITY:
Inclusion Criteria:

* patients met the definition of the Rome III criteria for FD

Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with functional dyspepsia primary care clinic were studied
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2010-10; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Estimated)

PRIMARY OUTCOMES:
Improvement of gastrointestinal Symptom as efficacy and the Number of Participants with Adverse Events as a Measure of Safety | 14 days

SECONDARY OUTCOMES:
Chinese version of the Nepean Dyspepsia Index as a Measure of efficacy | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Liu b yan, doctor, Study Director — Hunan university of TCM
Locations (1):
- Hunan university of TCM, Changsha, Hunan, China